CLINICAL TRIAL: NCT06585462
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 513 in Participants With Obesity
Brief Title: Single and Multiple Ascending Dose Study of AMG 513 in Participants With Obesity
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20230022
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cardiometabolic Disease
Keywords: AMG 513; Cardiometabolic disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (SAD) in Participants with Obesity (Part A) (Experimental): In Part A participants will enroll into SAD cohorts and will be randomized to receive AMG 513 or placebo subcutaneously (SC) or intravenously (IV).
  Interventions: Drug: AMG 513; Drug: Placebo
- Multiple Ascending Dose (MAD) in Participants with Overweight or Obesity (Part B) (Experimental): In Part B participants will enroll into MAD cohorts and will be randomized to receive AMG 513 or placebo SC.
  Interventions: Drug: AMG 513; Drug: Placebo

INTERVENTIONS:
Drug: AMG 513 — AMG 513 will be administered by SC or IV injection.
  Arms: Single Ascending Dose (SAD) in Participants with Obesity (Part A)
Drug: Placebo — Placebo will be administered by SC or IV injection.
  Arms: Single Ascending Dose (SAD) in Participants with Obesity (Part A)
Drug: AMG 513 — AMG 513 will be administered by SC injection.
  Arms: Multiple Ascending Dose (MAD) in Participants with Overweight or Obesity (Part B)
Drug: Placebo — Placebo will be administered by SC injection.
  Arms: Multiple Ascending Dose (MAD) in Participants with Overweight or Obesity (Part B)

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of AMG 513 after single and multiple doses.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the study will be males and females 18 to 65 years of age at the time of signing the informed consent with a body mass index (BMI) of 30.0 kg/m^2 to 40.0 kg/m^2 for Part A and BMI of 27.0 kg/m^2 to 40.0 kg/m^2 for Part B.
* Females enrolled must be of non-childbearing potential.

Exclusion Criteria:

* History and/or clinical evidence of diabetes mellitus, including hemoglobin A1c ≥ 6.5% and/or a fasting glucose of ≥ 126 mg/dL (7 mmol/L) at screening.
* Triglycerides ≥ 5.65 mmol/L (i.e., 500 mg/dL) at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-07-22 (Estimated); Study Completion 2026-07-22 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAE) | Approximately 178 days (Part A) and 225 days (Part B)

SECONDARY OUTCOMES:
Maximum Observed Drug Concentration (Cmax) of AMG 513 | Day 1 up to Day 57
Time to Cmax (Tmax) of AMG 513 | Day 1 up to Day 57
Area Under the Concentration-time Curve (AUC) of AMG 513 | Day 1 up to Day 57

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- United States (5):
  - Anaheim Clinical Trials, Anaheim, California
  - Orange County Research Center, Lake Forest, California
  - Fomat Medical Research, Oxnard, California
  - Translational Clinical Research LLC, Aventura, Florida
  - Clinical Pharmacology of Miami, LLC, Miami, Florida

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com